CLINICAL TRIAL: NCT03597633
Title: Tenofovir-based Combination Therapy or Monotherapy for Multi-drug Resistant Chronic Hepatitis B; Real World Data From Multicenter Cohort Study
Brief Title: Tenofovir Combination or Mono-therapy for MDR CHB
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Korea University (Other)
Collaborators: Yonsei University (Other); CHA University (Other); Soon Chun Hyang University (Other); Chonbuk National University (Other); Hallym University (Other); Inje University (Other); The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Hyung Joon Yim, Professor, Korea University
Other Study IDs: MDRCHB
Record Dates: First submitted 2018-07-16; First posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Chronic Hepatitis b With Multidrug Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Treatment of multidrug resistant (MDR) chronic hepatitis B (CHB) is still a challenging issue. Hence, the investigators will perform a multicenter prospective cohort study for the evaluation of tenofovir disoproxil fumarate (TDF)-based therapy for MDR CHB at real life settings.

DETAILED DESCRIPTION:
Inclusion criteria were CHB patients with resistance to more than two classes of nucleos(t)ide analogues (NA) and hepatitis B virus (HBV) DNA level ≥200 IU/mL.

Patients will receive either TDF-base combination therapy or TDF monotherapy. The primary end point is virologic response (VR) defined by an undetectable HBV DNA (<20 IU/mL) at month 36.

ELIGIBILITY:
Inclusion Criteria:

* CHB patients with:

  1. documented HBsAg positivity at least 6 months before enrollment
  2. age >18 years old,
  3. confirmed genotypic resistance to more than two classes of NAs
  4. HBV DNA level ≥ 200 IU/mL
  5. compensated liver diseases (defined by Child-Pugh-Turcotte score <7; prothrombin time <3 seconds above upper limit of normal or international normalized ratio <1.5; serum albumin >3 g/dL; total bilirubin <2.5 mg/dL; no history of esophago-gastric variceal bleeding, ascites, over hepatic encephalopathy)
  6. willingness to give an informed consent.

Exclusion Criteria:

1. laboratory abnormalities of low serum phosphorous level <2.0 mEq/dL, elevated serum creatinine >1.5 mg/dL, decreased creatinine clearance rate <50 mL/min, absolute neutrophil count <1000 cell/mL, or low hemoglobin level <10 g/dL (if female, <9 g/dL)
2. no definite evidence of genotypic resistance
3. positive antibody test for hepatitis C virus, hepatitis D virus, or human immunodeficiency virus
4. HCC
5. a proof of pregnant or lactating women
6. evidence of active alcohol consumption (140 g per a week for men and 70 g per a week for women)
7. any untreated malignancy.

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Chronic hepatitis B patients with multiple drug resistance.
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Virologic Response | 36 months
  undetectable HBV DNA (<20 IU/mL)

SECONDARY OUTCOMES:
Virologic Response | 60 months
  undetectable HBV DNA (<20 IU/mL)
mean HBV DNA | 36 months, 60 months
  mean HBV DNA levels
ALT normalization | 36 months, 60 months
  rates of ALT normalization
Hepatitis B e antigen (HBeAg) seroconversion | 36 months, 60 months
  rates of Hepatitis B e antigen (HBeAg) seroconversion
virologic breakthrough | 36 months, 60 months
  Incidence of virologic breakthrough defined by increase of HBV DNA more than 1 log IU/mL from nar dir.
Genotypic resistance | 36 months, 60 months
  Detection of previously known mutations to be resistant to the drugs being administered.

OTHER OUTCOMES:
Adverse event | 36 months, 60 months
  Any untoward event related or not related to the study medication

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Ansan Hospital, Ansan, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
Confidential